CLINICAL TRIAL: NCT01205009
Title: Human Chorionic Gonadotropin Supplementation Prior to In-vitro Fertilization Treatment in Poor Responders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Arik Tzukert, Hadassah Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hCGpoorresp-HMO-CTIL
Record Dates: First submitted 2010-08-30; First posted 2010-09-20 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2010-09

CONDITIONS: Infertility
Keywords: in-vitro fertilization; poor responders; human chorionic gonadotropin; Fertility Agents, Female
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

ARMS (2):
- Ovitrelle supplemantation (Active Comparator): The women will be given 250 mcg of Ovitrelle prior to their IVF cycle
  Interventions: Drug: Ovitrelle
- no Ovitrelle supplementation (No Intervention)

INTERVENTIONS:
Drug: Ovitrelle — One dose of Ovitrelle 250 mcg
  Arms: Ovitrelle supplemantation

SUMMARY:
In an era of delayed fertility plans, there is increasing need for fertility treatment in older women with poor response. Human chorionic gonadotropin (hCG) supplementation prior to treatment, as a thecal stimulant, may improve folliculogenesis and ovarian response.

ELIGIBILITY:
Inclusion Criteria:

* women >39 years on IVF treatment

Exclusion Criteria:

* polycystic ovary syndrome
* Any allergy to injection of human chorionic gonadotropin before

Ages: 40 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
number of oocytes retrieved | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mushira Aboo Dia, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel, Israel